CLINICAL TRIAL: NCT04622891
Title: Efficacy of Clarithromycin in Comparison to Azithromycin in Treatment of Mild COVID-19 Infection, Randomized Controlled Trial
Brief Title: Clarithromycin Versus Azithromycin in Treatment of Mild COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Alaa Rashad, Associate professor of chest diseases, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU-MED-CHT019-420860
Record Dates: First submitted 2020-11-06; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Covid19
Keywords: Azithromycin; clarithromycin; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Clarithromycin; Exercise; Azithromycin; Control Groups

STUDY DESIGN:
Intervention Model Description: clarithomycin group Azithromycin group control group
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- clarithromycin (Experimental): clarithromycin group
  Interventions: Drug: Clarithromycin 500mg
- Azithromycin (Active Comparator): azithromycin group
  Interventions: Drug: Azithromycin
- control (Placebo Comparator): control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clarithromycin 500mg — clarithromycin 500
  Other Names: active
  Arms: clarithromycin
Drug: Azithromycin — azithromycin group
  Other Names: active comparison
  Arms: Azithromycin
Drug: Placebo — control group
  Other Names: control group
  Arms: control

SUMMARY:
The current study was conducted at Qena Governorate, Egypt, during the period from May 2020, to July 2020. The study included 305 COVID-19 cases diagnosed by PCR, patients were randomly assigned to one of three study limps, Azithromycin 500 mg/24 h for 7 days, Clarithromycin 500 /12 h for 7 days, or a control group with no antibiotics, All three groups received only symptomatic treatment for control of fever and cough

DETAILED DESCRIPTION:
The current study was conducted at Qena Governorate, Egypt, during the period from May 2020, to July 2020. The study included 305 COVID-19 cases diagnosed by PCR, patients were randomly assigned to one of three study limps, Azithromycin 500 mg/24 h for 7 days, Clarithromycin 500 /12 h for 7 days, or a control group with no antibiotics, All three groups received only symptomatic treatment for control of fever and cough.

All study participants underwent full clinical evaluation including duration of fever, cough, dyspnea, anosmia or GIT symptoms, C-reactive protein (CRP), serum ferritin, D-dimer, Complete blood count (CBC), non-contrast chest computed tomography (CT) which was repeated 2 weeks after the start of treatment.

The Azithromycin group included, 107 patients, mean age 45.8 ±18 years, 73 male and 34 female, the Clarithromycin group included 99 patients mean age 46.1±19 years, 68 males and 31 female, the control group included 99 patients, with mean age 41.1 ± 18 years, 73 male and 28 female.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 cases
* Oxygen saturation > 93%
* Age >18 years

Exclusion Criteria:

* Patients <18 years,
* patients with Oxygen saturation < 93%, patients with
* Diabetes mellitus or
* heart failure,
* patients on chemotherapy or immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
time to fever control | 15 days
  time to complete resolution of fever

SECONDARY OUTCOMES:
PCR conversion | 15 days
  time to PCR conversion from first positive PCR for COVID-19 to negative PCR

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Rashad, MD, Principal Investigator — associate professor
Locations (1):
- south-Vally University faculty of medicine, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rashad A, Nafady A, Hassan MH, Mansour H, Taya U, Bazeed SES, Aref ZF, Sayed MAA, Nafady-Hego H, Abdelmaksoud AA. Therapeutic efficacy of macrolides in management of patients with mild COVID-19. Sci Rep. 2021 Aug 11;11(1):16361. doi: 10.1038/s41598-021-95900-z. PMID 34381155